CLINICAL TRIAL: NCT06741293
Title: Improving Colorectal Cancer Early Screening in Portugal: Identification and Validation of Biomarkers of Gut Microbiome in Stool
Brief Title: Improving Colorectal Cancer Early Screening in Portugal: Identification of Gut Microbiome Biomarkers in Stool (GUTBIOME-PT)
Acronym: GUTBIOME-PT
Status: Recruiting | Type: Observational
Sponsor: Gulbenkian Institute for Molecular Medicine (Other)
Collaborators: Hospital CUF Descobertas, Lisbon, Portugal (Unknown); CUF Tejo Hospital (Unknown); Hospital da Luz Lisboa, Portugal (Unknown)
Responsible Party: Sponsor
Other Study IDs: CAML Ref Nº: 111/23; 101060102 (Other Grant/Funding Number: European Union)
Record Dates: First submitted 2024-12-10; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer Screening; Colorectal Cancer (CRC); Microbiome
Keywords: colorectal cancer; microbiome; colorectal cancer screening; biomarkers; metagenomics
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Faecal samples with DNA - Participants will self-collect stool samples using a home collection kit into two tubes: one for FIT testing and the other for microbiome sequencing. Stool samples will be transported to the laboratory within 48 hours. FIT testing will be performed on its designated stool sample, while the samples for faecal microbiome sequencing will be subdivided into aliquots and stored at -80°C for subsequent shotgun metagenomics analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Control group: Healthy participants with a negative colonoscopy result
  Interventions: Other: No intervention: observational study
- Colorectal cancer: Participants with colorectal cancer diagnosis confirmed by colonoscopy
  Interventions: Other: No intervention: observational study
- Low-risk polyps: Participants with positive colonoscopy and detection of low-risk adenomas
  Interventions: Other: No intervention: observational study
- High-risk polyps: Participants with positive colonoscopy and detection of high-risk adenomas
  Interventions: Other: No intervention: observational study

INTERVENTIONS:
Other: No intervention: observational study — No intervention: observational study

SUMMARY:
Colorectal cancer (CRC) is a major public health problem, responsible for 2 million new cases and almost 1 million deaths annually worldwide. In Portugal, as of 2022, CRC is the most common cancer, with 10,575 new cases reported, and the second leading cause of cancer-related mortality, accounting for 4,809 deaths (approximately 14% of all cancer-related deaths). In recent years, there has been an alarming increase in the incidence and mortality of CRC in people <50 years of age.

Early detection is crucial, as survival rates decline sharply from 90% when detected early to just 10% in advanced stages. Non-invasive diagnostic tests, such as the Faecal Immunochemical Test (FIT), have a low sensitivity for early-stage lesions and a high rate of false positives. Therefore, there is an urgent need to improve non-invasive diagnostic methods for the early detection of CRC, as effective screening can prevent it by detecting and removing premalignant lesions.

Recent studies suggest that an altered gut microbiota may confer susceptibility to certain types of cancer. Interestingly, the gut microbiota of patients with adenomas or CRC differs from that of healthy individuals. This study aims to identify gut microbiome biomarkers in faecal samples associated with CRC and/or high-risk adenomas to improve early detection.

DETAILED DESCRIPTION:
This study will analyse the gut microbiome in stool samples collected from individuals living in the Lisbon Metropolitan Area, Portugal. Using shotgun metagenomics, the investigators aim to identify microbiome biomarkers associated with the early detection of CRC and the progression of precancerous lesions (adenomas). The identified biomarkers will be tested to develop a non-invasive and highly sensitive screening tool for CRC and precancerous lesions.

Primary Objective:

To identify gut microbiome biomarkers in faecal DNA associated with CRC and/or high-risk adenomas.

Secondary Objectives:

i) Establish the correlation between FIT results, faecal microbiome testing and colonoscopy results.

ii) Estimate the incidence of CRC in the Lisbon Metropolitan Area among individuals aged 40-74 years, stratified by sex and age group.

iii) Analyse associations between clinical data (e.g., clinical history, lifestyle, and dietary habits), faecal microbiome profiles, FIT results, and colonoscopy outcomes, comparing individuals with CRC and/or high-risk adenomas against healthy individuals, for the total sample and by sex and age group; iv) Identify risk factors (e.g., clinical history, lifestyle, dietary habits) associated with CRC development, stratified by sex and age group.

Study Design:

This is an observational, prospective, longitudinal study involving individuals aged 40-74 years residing in the Lisbon Metropolitan Area who voluntarily enrol in the study.

Participants meeting all inclusion criteria and no exclusion criteria (as detailed in the relevant section) will be included. Based on sample size calculations using the Neyman allocation formula and taking as a reference the distribution of the population living in the Lisbon Metropolitan Area (stratified by sex and age groups: 40-49, 50-59, 60-64, 65-69 and 70-74 years), along with assumptions of the overall FIT test prevalence and sensitivity, a total of 30.000 participants will be enrolled.

At baseline, participants will provide a faecal sample within 2 to 10 days of enrolment. Demographic, clinical, and lifestyle data-including age, family history of CRC, personal medical history, smoking habits, physical activity levels, stress, and body mass index (BMI)-will be collected via self-administered questionnaires. Dietary habits and adherence to the Mediterranean diet will be assessed through telephone interviews.

Participants will be followed for six years, with faecal samples collected every 2 years. Clinical and lifestyle data will also be updated every two years throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study procedures
* Reside in the Lisbon Metropolitan Area,, Portugal
* Age from 40 to 74 years

Exclusion Criteria:

* Age < 40 years or ≥ 75 years
* Unable to provide informed consent
* Refusal to provide stool samples
* Active oncological disease
* Personal history of CRC
* Personal history of colon adenomas removed in the last 24 months
* First-degree family history of CRC
* Previous diagnosis of inflammatory bowel disease (ulcerative colitis, Crohn's disease or indeterminate colitis), inflammatory bowel syndrome, persistent and infectious gastroenteritis, colitis or gastritis, persistent or chronic diarrhoea of unknown aetiology or recurrent infection by Clostridioides difficile
* Severe cardiovascular or heart diseases with medical diagnosis
* Severe renal failure requiring hemodialysis
* Severe lung disease
* Pregnancy

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two different recruiting strategies will be used:
  * Opportunistic recruitment: recruitment will be conducted in collaboration with the gastroenterology and general medicine departments of partner hospitals in Lisbon. Eligible individuals scheduled for a screening colonoscopy will be informed about the study by an on-site study coordinator. Those willing to participate will sign an informed consent form.
  * Random recruitment: interested individuals can access detailed information and assess their eligibility by completing an online questionnaire on the study's website. Eligible participants can register and provide informed consent digitally. After registration, participants will be contacted to arrange the delivery of a self-collection kit for stool sample collection.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2025-11-28 (Estimated); Study Completion 2029-11-28 (Estimated)

PRIMARY OUTCOMES:
Microbiome biomarkers associated with CRC and/or high-risk polyps. | Baseline and Follow-up every 2 years up to 6 years
  The faecal microbiota composition and gene profiles will be analysed using shotgun metagenomic sequencing on a subset of participants (up to 10,000 samples). Data will be integrated with lifestyle, dietary factors and colonoscopy results to identify biomarkers linked to CRC and adenomas.
Correlation between microbiome biomarkers and FIT results | Baseline and Follow-up every 2 years up to 6 years
  Faecal microbiome analysis results will be compared with FIT test results to evaluate the predictive value, negative predictive value, and overall effectiveness in detecting CRC in an asymptomatic population.

SECONDARY OUTCOMES:
Effect of diet on CRC risk and gut microbiota composition | Baseline
  Dietary intake will be assessed via telephone interview through two 24-hour recalls, following the protocol validated by the European Food Safety Authority (EFSA).
Effect of the Mediterranean Diet on CRC risk and gut microbiota composition | Baseline
  Adherence to the Mediterranean Diet will be assessed using the PREvención con DIeta MEDiterránea (PREDIMED) nutritional questionnaire, a validated 14-item tool. Each question is scored either 0 (condition not met) or 1 (condition met), resulting in a total score ranging from 0 to 14 (7). Based on this final score, adherence to the Mediterranean Diet will then be categorised into three groups: low adherence (score < 5), moderate adherence (score 6-9), and high adherence (score > 10)
Effect of physical activity on CRC risk and gut microbiota composition | Baseline
  Physical activity will be assessed using the Nordic Physical Activity Questionnaire-short form, a validated tool composed of two close-ended questions for monitoring adherence to WHO physical activity recommendations. Participants will be categorized as "Below WHO physical activity recommendations" or "Equal to WHO physical activity recommendations"
Effect of sleeping habits on CRC risk and gut microbiota composition | Baseline
  Sleeping habits will be assessed by the Pittsburgh Sleep Quality Index (PSQI), a validated questionnaire that consists of 19 items which are distributed into seven "components": subjective sleep quality; sleep latency; sleep duration; habitual sleep efficiency; sleep disturbances; use of sleeping medication; day-time dysfunction. Each component is scored from 0 a 2, and the sum of the component scores yields a global PSQI score. A global PSQI score ≥6 will indicate poor sleep quality.
Effect of stress levels on CRC risk and gut microbiota composition | Baseline
  Stress levels will be assessed by the Perceived Stress Scale, a validated questionnaire composed of 10 questions. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 will be considered low stress, 14-26 will be considered moderate stress and scores ranging from 27-40 will be considered high perceived stress.
Risk factors (medical history, lifestyle and dietary habits) associated with CRC and/or high-risk polyps | Baseline and Follow-up every 2 years up to 6 years
  Eligible participants will be invited to participate every two years over six years. Longitudinal data will identify significant risk factors for the development of CRC or high-risk polyps.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulbenkian Institute for Molecular Medicine, Lisbon, Lisbon District, Portugal

REFERENCES:
- See also: Public study website — https://www.nodabarriga.pt/Homepage